CLINICAL TRIAL: NCT06889441
Title: Effect of Pacifier Use on Motor Development and Sensory Processing Skills in Infants
Brief Title: Pacifier Use and Infant Development
Status: Completed | Type: Observational
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Rabia ZORLULAR, principal investigator, Nigde Omer Halisdemir University
Other Study IDs: pacifier use
Record Dates: First submitted 2025-03-15; First posted 2025-03-21 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-03

CONDITIONS: Pacifier; Infant Development; Sensory Processing Disorder
Keywords: Pacifier use; development; Sensory Processing Skills; motor development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- pacifier user: Full-term infants who have used a pacifier for at least 6 months will be included in the study. The infants' motor development and sensory processing skills will be evaluated.
  Interventions: Behavioral: Test of sensory function in infants; Behavioral: The Peabody Developmental Motor Scales-Second Edition; Behavioral: Infant/toddler sensory profile
- non-pacifier: The motor development and sensory processing skills of full-term infants who are 9-12 months old and do not use a pacifier will be evaluated. The developmental results of both groups will be compared
  Interventions: Behavioral: Test of sensory function in infants; Behavioral: The Peabody Developmental Motor Scales-Second Edition; Behavioral: Infant/toddler sensory profile

INTERVENTIONS:
Behavioral: Test of sensory function in infants — It was planned to use the Test of sensory function in infants to evaluate the sensory development of infants. The test of sensory function in infants is frequently used to evaluate the sensory processing functions of infants aged 4-18 months. It is used to determine whether an infant has a sensory processing problem and to what extent. It consists of 24 items. The test of sensory function in infants requires the infant to be stimulated and interacted with various materials. The total score varies between 0-49 and the test has normative values for different age groups. Although it is used from the fourth month onwards, the most reliable and valid results are obtained between 7-18 months.
Behavioral: The Peabody Developmental Motor Scales-Second Edition — The Peabody Developmental Motor Scales-Second Edition is a standardized, norm-referenced assessment instrument designed to evaluate both gross and fine motor skills in children aged 0 to 71 months. It is frequently employed in clinical, educational, and research contexts to detect motor developmental delays, monitor developmental trajectories, and inform intervention strategies. Notably, higher scores on the scale reflect superior motor performance, indicating better developmental outcomes
Behavioral: Infant/toddler sensory profile — The infant/toddler sensory profile is a questionnaire filled out by the child's primary caregiver to collect information about sensory processing abilities. The test evaluates sensory processing in 6 different areas. These items consist of general, visual, auditory, vestibular, tactile and oral sensory processing. The caregiver evaluates the child's behavior on a 5-point scale. One point means "almost always" and five points means "almost never". The caregiver's responses are summarized using standard scoring procedures and then interpreted in terms of the impact of a child's sensory processing abilities on the child and their family's lives. The scores are normative for age and are important in assessing sensory development.

SUMMARY:
Pacifier use reduces the risk of sudden infant death syndrome, and nonnutritive sucking has been shown to improve physiological balance and feeding in premature infants. Therefore, the risks and benefits of pacifier use should be carefully considered. In a study, it was reported that giving a pacifier on the 15th day did not change the prevalence and duration of breastfeeding, that using a pacifier was associated with a lower incidence of sudden infant death syndrome, and that giving a pacifier was a useful approach. Using a pacifier can help the baby calm down and adapt to the environment. When the literature was reviewed, conflicting results were reported regarding using a pacifier. However, the effect of using a pacifier on the baby's motor development and especially sensory processing skills has not been clearly investigated.

DETAILED DESCRIPTION:
Pacifier use is a very common practice. It is often used in the early years of a child's life to help them fall asleep or to soothe and calm them down from teething pain. The age at which a pacifier is discontinued is usually around the age of three when the child goes to nursery. Observational studies have linked early pacifier use with breastfeeding problems leading to early weaning. However, randomized controlled trials have not shown a similar negative association between early pacifier use and successful breastfeeding, suggesting that pacifier use may be a sign of breastfeeding problems and not the cause. Pacifier use is often a topic of debate when parents and professionals aim to maintain and support breastfeeding. However, the literature supports the beneficial effects of pacifier use in infants because of the associated physiological benefits, such as digestion, behavioral organization, pain management, motor function, and sucking development.

Pacifier use reduces the risk of sudden infant death syndrome, and nonnutritive sucking has been shown to improve physiological balance and feeding in premature infants. Therefore, the risks and benefits of pacifier use should be carefully considered. In a study, it was reported that giving a pacifier on the 15th day did not change the prevalence and duration of breastfeeding, that using a pacifier was associated with a lower incidence of sudden infant death syndrome, and that giving a pacifier was a useful approach. Using a pacifier can help the baby calm down and adapt to the environment. When the literature was reviewed, conflicting results were reported regarding using a pacifier. However, the effect of using a pacifier on the baby's motor development and especially sensory processing skills has not been clearly investigated. The aim of this study was to evaluate babies using a pacifier in terms of both motor development and sensory processing skills and to compare them with their peers who did not use a pacifier.

ELIGIBILITY:
Inclusion Criteria:

* Full-term infants who have used a pacifier for at least 6 months and are still using it,
* Babies who do not have sucking dysfunction and are breastfed for the first 6 months,
* Post-term infants who are between 9-12 months old

Exclusion Criteria:

* Premature infants
* Infants with congenital malformations
* Infants diagnosed with metabolic, neurological and genetic diseases
* Children whose parents do not volunteer for the study

Ages: 9 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Full-term infants who have used a pacifier for at least 6 months and full-term infants who have never used a pacifier will be included in the study. The motor and sensory development of the included children will be compared according to their pacifier use status.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2025-03-21 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Peabody Developmental Motor Scales | Second Edition | 9-12 months
  The Peabody Developmental Motor Scales-Second Edition is a standardized, norm-referenced assessment instrument designed to evaluate both gross and fine motor skills in children aged 0 to 71 months. The Peabody Developmental Motor Scales-Second Edition comprises six subtests, namely Reflexes, Stationary, Locomotion, Object Manipulation, Grasping, and Visual-Motor Integration, which collectively measure a broad spectrum of motor functions including postural control, locomotor abilities, object manipulation, and hand-eye coordination. The subtests generate three composite scores: the Gross Motor Quotient, Fine Motor Quotient, and Total Motor Quotient, offering a comprehensive evaluation of a child's motor competence. Notably, higher scores on the scale reflect superior motor performance, indicating better developmental outcomes
Test of Sensory Functions in Infants | 9-12 months
  It was planned to use the Test of sensory function in infants to evaluate the sensory development of infants. The test of sensory function in infants is frequently used to evaluate the sensory processing functions of infants aged 4-18 months. It is used to determine whether an infant has a sensory processing problem and to what extent. It consists of 24 items. The test of sensory function in infants requires the infant to be stimulated and interacted with various materials. The total score varies between 0-49 and the test has normative values for different age groups. Although it is used from the fourth month onwards, the most reliable and valid results are obtained between 7-18 months.
Infant/toddler sensory profile | 9-12 months
  Infant/toddler sensory profile; The infant/toddler sensory profile is a questionnaire filled out by the child's primary caregiver to collect information about sensory processing abilities. It is a questionnaire that questions the behavior and performance of a child between the ages of 0-3 (0-7 months and 7-36 months) regarding sensory processing. The test evaluates sensory processing in 6 different areas. These items consist of general, visual, auditory, vestibular, tactile and oral sensory processing. The caregiver evaluates the child's behavior on a 5-point scale. One point means "almost always" and five points means "almost never". The caregiver's responses are summarized using standard scoring procedures and then interpreted in terms of the impact of a child's sensory processing abilities on the child and their family's lives. The scores are normative for age and are important in assessing sensory development.

CONTACTS AND LOCATIONS:
Overall Officials: Rabia ZORLULAR, Principal Investigator — Nigde Omer Halisdemir University
Locations (1):
- Nigde Omer Halisdemir University, Niğde, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cabral TI, Pereira da Silva LG, Tudella E, Simoes Martinez CM. Motor development and sensory processing: A comparative study between preterm and term infants. Res Dev Disabil. 2015 Jan;36C:102-107. doi: 10.1016/j.ridd.2014.09.018. Epub 2014 Oct 16. PMID 25462470
- [Background] Dunn, W. and D.B. Daniels, Initial development of the infant/toddler sensory profile. Journal of Early Intervention, 2002. 25(1): p. 27-41.
- [Background] Howard CR, Howard FM, Lanphear B, Eberly S, deBlieck EA, Oakes D, Lawrence RA. Randomized clinical trial of pacifier use and bottle-feeding or cupfeeding and their effect on breastfeeding. Pediatrics. 2003 Mar;111(3):511-8. doi: 10.1542/peds.111.3.511. PMID 12612229
- [Background] Barnes DM, Hanby AM, Gillett CE, Mohammed S, Hodgson S, Bobrow LG, Leigh IM, Purkis T, MacGeoch C, Spurr NK, et al. Abnormal expression of wild type p53 protein in normal cells of a cancer family patient. Lancet. 1992 Aug 1;340(8814):259-63. doi: 10.1016/0140-6736(92)92354-i. PMID 1353190